CLINICAL TRIAL: NCT03213704
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of LOXO-101 (Larotrectinib) in Patients With Tumors Harboring Actionable NTRK Fusions
Brief Title: Larotrectinib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With NTRK Fusions (A Pediatric MATCH Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01264; NCI-2017-01264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621A; APEC1621A (Other: Children's Oncology Group); APEC1621A (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Ependymoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Kidney Wilms Tumor; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Glioma; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Refractory Ependymoma; Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Refractory Glioma; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Primary Central Nervous System Neoplasm; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma
MeSH Terms: conditions — Ependymoma; Neuroectodermal Tumors, Primitive, Peripheral; Glioma; Hepatoblastoma; Wilms Tumor; Histiocytosis, Langerhans-Cell; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Central Nervous System Neoplasms | interventions — Specimen Handling; Biopsy; larotrectinib; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (larotrectinib sulfate) (Experimental): Patients receive larotrectinib sulfate PO or via NG- or G-tube BID on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, MRI, an x-ray, bone scan, and/or MIBG scintigraphy during screening and on study. Patients also undergo bone marrow aspiration and/or biopsy during screening and may undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Larotrectinib Sulfate; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow aspiration and/or biopsy
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Larotrectinib Sulfate — Given PO or via nasogastric- or gastric-tube
  Other Names: ARRY 470 Sulfate; LOXO 101 Sulfate; LOXO-101 Sulfate; Vitrakvi
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Radionuclide Imaging — Undergo a MIBG scintigraphy
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II Pediatric MATCH trial studies how well larotrectinib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with NTRK fusions that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and have come back (relapased) or does not respond to treatment (refractory). Larotrectinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with larotrectinib sulfate (LOXO-101 [larotrectinib]) with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders harboring NTRK 1/2/3 fusions.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with LOXO-101 (larotrectinib) with advanced solid tumors (including CNS tumors), non-Hodgkin lymphomas or histiocytic disorders with NTRK 1/2/3 fusions.

II. To obtain additional information about the tolerability of LOXO-101 (larotrectinib) in children with relapsed or refractory cancer.

III. To provide preliminary estimates of the pharmacokinetics of LOXO-101 (larotrectinib) in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVE:

I. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive larotrectinib sulfate orally (PO) or via nasogastric (NG)- or gastric (G)-tube twice per day (BID) on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a computed tomography (CT) scan, magnetic resonance imaging (MRI), an x-ray, bone scan, and/or iobenguane (MIBG) scintigraphy during screening and on study. Patients also undergo bone marrow aspiration and/or biopsy during screening and may undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days, then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* APEC1621SC: Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621A based on the presence of an actionable mutation as defined in APEC1621SC
* Patients must be >= than 12 months and =< 21 years of age at the time of study enrollment
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have MIBG+ evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard MRI or CT; Note: The following do not qualify as measurable disease:

  * Malignant fluid collections (e.g., ascites, pleural effusions)
  * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
  * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
  * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
  * Previously radiated lesions that have not demonstrated clear progression post radiation
  * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required time frame, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; for agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil [ANC] counts): >= 7 days after the last dose of agent; for agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor leukocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, NK cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial brain metastases (BM) radiation; Note: radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to other NTRK inhibitors including but not limited to LOXO-101 (larotrectinib), entrectinib (RXDX-101), DS6051, PLX7486
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment)
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (within 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 (within 7 days prior to enrollment) or
* A serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL); male: 0.6 female: 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL); male: 0.8 female: 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL); male: 1 female: 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL); male: 1.2 female: 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL); male: 1.5 female: 1.4
  * Age: >= 16 years; maximum serum creatinine (mg/dL); male: 1.7 female: 1.4
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment); (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Patients with seizure disorder may be enrolled if on anti-convulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflect (DTR); any grade of DTR is eligible
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study treatment
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease (GVHD) post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible; strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study; Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
* Patients who have received prior therapy with a specific inhibitor of TRK (including but not limited to entrectinib [RXDX-101], DS-6051b, and PLX7486) are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-10-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Janeway, Principal Investigator — Children's Oncology Group
Locations (124):
- United States (122):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Larotrectinib Sulfate)
Started | 9
Completed | 1
Not Completed | 8
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1
Not completed — Progressive disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Larotrectinib Sulfate)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors).
Time Frame: Up to 2 years from study entry
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Larotrectinib Sulfate)
Number analyzed (Participants) | 9
percentage of participants | 33 [14.2 to 60.2]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 6 month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact.
Time Frame: Up to 6 months from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Larotrectinib Sulfate)
Number analyzed (Participants) | 9
percentage of participants | 76 [33.2 to 93.5]

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or Higher Adverse Events
Description: Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 2 years from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Larotrectinib Sulfate)
Number analyzed (Participants) | 9
percentage of participants | 44 [13.7 to 78.8]

4. Other Pre Specified Outcome: Pharmacokinetics of Larotrectinib
Description: A descriptive analysis of pharmacokinetic parameters of LOXO-101 (larotrectinib) will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The pharmacokinetic parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit). All these analyses will be descriptive and exploratory and hypotheses generating in nature.
Time Frame: Pre-dose, 1, 2, 4, and 6-8 hours after morning dose of day 1 cycle 1 and pre-dose of day 1 cycle 2
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Ability to Detect NTRK Fusions in Circulating Cell-free Tumor Deoxyribonucleic Acid in Plasma
Description: A descriptive analysis of the exploratory aims will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment to 30 days after the end of treatment, up to 2 years. All-Cause Mortality monitored/assessed up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Larotrectinib Sulfate)
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Larotrectinib Sulfate) (N=9)
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Fever (General disorders) | 1
Sepsis (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Larotrectinib Sulfate) (N=9)
Anemia (Blood and lymphatic system disorders) | 4
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 1
Scleral disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Localized edema (General disorders) | 1
Pain (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Otitis media (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Hemoglobin increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 3
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03213704/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03213704/ICF_001.pdf